CLINICAL TRIAL: NCT05820269
Title: InterventionPredictive Factors for the Outcome of Emotional and/or Behavioural Disorders in 18- to 48 Month-old Children After Psychotherapeutic Intervention
Brief Title: Predictive Factors for the Outcome of Young Children Emotional and/or Behavioral Disorders After Psychotherapeutic Intervention
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 8301
Record Dates: First submitted 2023-03-22; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Behavioral Disorders; Emotional Disorder of Childhood
Keywords: childhood; Behavioral Disorders; Emotional Disorder of Childhood
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: parents-child psychotherapy — filling out questionnaires during psychotherapy consultations

SUMMARY:
Behavioral disorders and emotional disorders represent frequent reasons for consultation in young children.

Their prevalence is between 7% and 13% depending on the studies. Behavioral disorders, and to a lesser extent emotional disorders, tend to persist through childhood and adolescence and are a risk factor for disorders in adulthood.

There is still little research on psychotherapies concerning children and even less on parent(s)-young child therapies, despite a certain interest of clinicians for these.

In a previous study, three independent factors appeared predictive of the unfavorable child's outcome : the frequency and intensity of behavioral problems and fears, as well as the absence of the father at more than 2/3 of the consultations. The only independent factor associated with the outcome of the mother was her anxiety score at the start of treatment.

The study presented here will take these elements into account and will include an assessment of both parents.

The main objective is to identify predictive factors of behavioural and emotional disorder outcome in children aged 18 months to 48 months after parent-child psychotherapy. The secondary objectives are to study predictive factors of the outcome in parents (anxiety/depression symptoms) and parent-child relationship.

The main predictive factors will be the presence of the father at the consultations, the therapeutic alliance (subject to validation), the type of disorder of the child and the parental psychopathology.

DETAILED DESCRIPTION:
Behavioral disorders and emotional disorders represent frequent reasons for consultation in young children.

Their prevalence is between 7% and 13% depending on the studies. Behavioral disorders, and to a lesser extent emotional disorders, tend to persist through childhood and adolescence and are a risk factor for disorders in adulthood.

There is still little research on psychotherapies concerning children and even less on parent(s)-young child therapies, despite a certain interest of clinicians for these.

Most studies have shown a significant association between these early childhood disorders and a parent-child relationship disorder, as well as the presence of depressive symptoms in the mother.

Other risk factors include environmental, child and parenting factors.

Several types of therapeutic intervention have been developed in recent decades to treat the difficulties of young children, their common point being to work jointly with the child and the parents and to focus on the parent-child relationship.

From the many studies carried out, we can retain the greatest difficulty in treating behavioral disorders, compared to emotional disorders or functional disorders.

Even if the therapies have shown their effectiveness, a certain number of children continue to present difficulties after the treatment.

The factors most often found associated with poorer progress are the intensity of the child's disorders, the child's advanced age, the presence of parental psychopathology and negative life events.

In young children, other studies are needed to better understand the factors involved in the failure or success of therapy and in particular to determine whether these are the same factors as in older children.

Several early childhood clinicians have insisted on the need for an alliance so that therapeutic work can take place. In particular, they underlined the importance of developing empathy and a positive affective bond between the therapist and the parents. Despite its recognized clinical interest, the therapeutic alliance (or working alliance) has been the subject of little research in populations of young children.

The "Working Alliance Inventory" is a scale measuring the therapeutic alliance differentiates three components: the bond, the tasks and the objectives

In a previous study, three independent factors appeared predictive of the unfavorable future of the child: the frequency and intensity of behavioral problems and fears, as well as the absence of the father at more than 2/3 of the consultations. The only independent factor associated with the outcome of the mother was her anxiety score at the start of treatment.

The study presented here will take these elements into account and will include an assessment of both parents.

The main objective is to identify predictive factors of behavioural and emotional disorder outcome in children aged 18 months to 48 months after parent-child psychotherapy. The main outcome is the Child Beavior Check list (CBCL) total score change.

The secondary objectives are to study predictive factors of the outcome in parents (anxiety/depression symptoms) and parent-child relationship.

Outcomes will be assessed by comparing the pre- and post-therapy scores of a battery of questionnaires that assess the child's symptoms, the parents' anxiety/depression, and the parent-child relationship. Multivariate linear regression analysis will be used to identify, among the studied variables (child age and sex, socio-economic status, life events, disorder type, intensity and duration, social support, parents' psychopathology, parents' attachment, parent-child relationships, therapy length and frequency, father's involvement in the therapy, and therapeutic alliance), predictive factors of the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* first medico-psychological consultation with a young child and one or both parents
* child aged 18 to 48 months at the time of making the appointment for the first consultation
* parents who can speak French
* child presenting as a reason for consultation a behavioral and/or a emotional disorder (anger, opposition, provocation, aggressiveness, hyperactivity, agitation, fits of crying, separation difficulties, exaggerated fears, anxiety, sadness, shyness, withdrawal)
* parents who signed the written consent
* affiliation to a social security scheme

Exclusion Criteria:

* child referred on therapeutic injunction by the judicial services
* child seen only for a diagnostic opinion, with redirection to another service or private for pick-up if needed
* presence of an adult other than the father or mother at the first consultation (apart from a mother-in-law or father-in-law)
* child with a suspected or diagnosed pervasive developmental disorder (according to ICD10, F84 criteria),
* suspicion or diagnosis of physical abuse
* child with a sensory disability or mental retardation already diagnosed
* child referred by a SESSAD, a CAMSP or an assessment center for pervasive disorders of the development

Ages: 18 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: child with behavioral problems or emotional disorders consulting in a psychological care service
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2009-01-05 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
predictive factors of behavioural disorder outcome | between inclusion and 18 months
  The evolution of the child will be the total score of the CBCL (a z-score < 1 will be considered as a favorable evolution).
predictive factors of emotional disorder outcome | between inclusion and 18 months
  Parent-child relationships will be calculated by the PIR-GAS score.
  Relationship difficulties are assessed based on the intensity, frequency and duration of maladaptive interactions and a score below 40 indicates a disordered relationship.

SECONDARY OUTCOMES:
predictive factors of the outcome in parents (anxiety/depression symptoms) and parent-child relationship | at 18 months
  validate the IT-WAI-S (Infant-Toddler Working Alliance Inventory short version, a therapeutic alliance assessment tool, translated in French from the Working alliance Inventory and adapted to early consultations

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Joëlle Hervé, PHD, Principal Investigator — UH of Montpellier
Locations (1):
- UH of Montpellier, Montpellier, France